CLINICAL TRIAL: NCT01344993
Title: A Phase I/II, Open-Label, Multi-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (MA09-hRPE) Cells in Patients With Advanced Dry AMD
Brief Title: Safety and Tolerability of Sub-retinal Transplantation of hESC Derived RPE (MA09-hRPE) Cells in Patients With Advanced Dry Age Related Macular Degeneration
Acronym: Dry AMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7316-CL-0002; ACT MA09-hRPE AMD-001 (Other: Sponsor)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Dry Age Related Macular Degeneration
Keywords: Dry AMD; Geographic atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MA09-hRPE (Experimental): Experimental: Subretinal injection of MA09-hRPE
  * Cohort 1 50,000 cells
  * Cohort 2 100,000 cells
  * Cohort 2a Better Vision 100,000 cells
  * Cohort 3 150,000 cells
  * Cohort 4 200,000 cells
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — Cohort 1 50,000 cells Cohort 2 100,000 cells Cohort 2a Better Vision 100,000 cells Cohort 3 150,000 cells Cohort 4 200,000 cells

SUMMARY:
This is a safety and tolerability trial to evaluate the effect of subretinal injection of human embryonic stem cell derived retinal pigment epithelium cells in patients with dry Age Related Macular Degeneration (AMD) and to perform exploratory evaluation of potential efficacy endpoints to be used in future studies retinal pigment epithelium (RPE) cellular therapy.

DETAILED DESCRIPTION:
This study is a Phase I/II, open-label, non randomized, sequential, multi-center clinical trial. There will be 5 cohorts, the 4 low vision cohorts will contain 3 patients, the better vision cohort will contain 4 patients. The enrolled cohorts will be as follows:

Three AMD patients- 50,000 MA09-hRPE cells transplanted Three AMD patients- 100,000 MA09-hRPE cells transplanted Four Better Vision AMD patients- 100,000 MA09-hRPE cells transplanted Three AMD patients- 150,000 MA09-hRPE cells transplanted Three AMD patients- 200,000 MA09-hRPE cells transplanted

Patients will be enrolled sequentially, and within each cohort of 3 patients, each patient's clinical course over the first 6 weeks following cell transplantation will be reviewed by an independent (DSMB) before enrollment is opened for the next 2 patients. A full safety assessment of all 3 patients in each cohort will be made by the DSMB when the 3rd patient in each cohort completes 4 weeks of follow-up, and before the first patient in the next cohort receives a cell transplant. The exception is the better vision group where all patients may be enrolled once DSMB approval has been received.

Each cohort will be enrolled sequentially in turn, with the exception of the better vision cohort which may be enrolled in parallel with the other cohorts.

The day of the cell implantation will be Day 0, and patients will remain in the study until the last visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female over 55 years of age.
* Patient should be in sufficiently good health to reasonably expect survival for at least four years after treatment
* Clinical findings consistent with advanced dry AMD with evidence of one or more areas of >250microns of geographic atrophy (as defined in the Age-Related eye Disease Study [AREDS] study) involving the central fovea.
* GA defined as attenuation or loss of RPE as observed by biomicroscopy, OCT, and FA.
* No evidence of current or prior choroidal neovascularization in the treated eye
* The visual acuity of the eye to receive the transplant will be no better than 20/400. The visual acuity of the eye in the better vision cohort to receive the transplant will be no better than 20/100.
* The visual acuity of the eye that is not to receive the transplant will be no better than 20/400 for the worse vision patients and no worse than 20/100 for the better vision patients.
* Electrophysiological findings consistent with advanced dry AMD.
* Medically suitable to undergo vitrectomy and subretinal injection.
* Medically suitable for general anesthesia or waking sedation, if needed.
* Medically suitable for transplantation of an embryonic stem cell line:

Any laboratory value which falls slightly outside of the normal range will be reviewed by the Medical Monitor and Investigators to determine its clinical significance. If it is determined not to be clinically significant, the patient may be enrolled into the study.

* Normal serum chemistry (sequential multi-channel analyzer 20 [SMA-20]) and hematology (complete blood count [CBC], prothrombin time [PT], and activated partial thromboplastin time [aPTT]) screening tests. (NOTE:With the exception of abnormalities specifically identified in the exclusion criteria)
* Negative urine screen for drugs of abuse.
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serologies.
* No history of malignancy (with the exception of successfully treated (excised) basal cell carcinoma[skin cancer] or successfully treated squamous cell carcinoma of the skin).
* Negative cancer screening within previous 6 months:
* complete history & physical examination;
* dermatological screening exam for malignant lesions;
* negative fecal occult blood test & negative colonoscopy within previous 7 years;
* negative chest roentgenogram (CXR);
* normal CBC & manual differential;
* negative urinalysis (U/A);
* normal thyroid exam;
* if male, normal testicular examination; digital rectal examination (DRE) and prostate specific antigen (PSA);
* if female, normal pelvic examination with Papanicolaou smear; and
* If female, normal clinical breast exam and, negative mammogram.
* If female and of childbearing potential, willing to use two effective forms of birth control during the study.
* If male, willing to use barrier and spermicidal contraception during the study.
* Willing to defer all future blood, blood component or tissue donation.
* Able to understand and willing to sign the informed consent

Exclusion Criteria:

* Presence of active or inactive CNV in the eye to be treated.
* Presence or history of retinal dystrophy, retinitis pigmentosa, chorioretinitis, central serious choroidopathy, diabetic retinopathy or other retinal vascular or degenerative disease other than ARMD.
* History of optic neuropathy.
* Macular atrophy due to causes other than AMD.
* Presence of glaucomatous optic neuropathy in the study eye, uncontrolled IOP, or use of two or more agents to control IOP (acetazolamide, beta blocker, alpha-1-agonist, antiprostaglandins, anhydrous carbonic inhibitors).
* Cataract of sufficient severity likely to necessitate surgical extraction within 1 year.
* History of retinal detachment repair in the study eye.
* Axial myopia of greater than -8 diopters
* Axial length greater than 28 mm.
* History of malignancy (with the exception of successfully treated [excised] basal cell carcinoma[skin cancer] or successfully treated squamous cell carcinoma of the skin).
* History of myocardial infarction in previous 12 months.
* History of diabetes mellitus.
* History of cognitive impairments or dementia which may impact the patients ability participate in the informed consent process and to appropriately complete evaluations.
* Any immunodeficiency.
* Any current immunosuppressive therapy other than intermittent or low dose corticosteroids.
* Alanine transaminase/aspartate aminotransferase (ALT/AST) >1.5 times the upper limit of normal or any known liver disease.
* Renal insufficiency, as defined by creatine level >1.3 mg/dL.
* A hemoglobin concentration of less than 10 gm/dL, a platelet count of less than 100k/mm3 or an absolute neutrophil count of less than 1000/mm3 at study entry.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV.
* Current participation in any other clinical trial.
* Participation within previous 6 months in any clinical trial of a drug by ocular or systemic administration.
* Any other sight-threatening ocular disease.
* Any history of retinal vascular disease (compromised blood-retinal barrier.
* Glaucoma.
* Uveitis or other intraocular inflammatory disease.
* Significant lens opacities or other media opacity.
* Ocular lens removal within previous 3 months.
* Ocular surgery in the study eye in the previous 3 months
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06-09 (Actual); Primary Completion 2015-08-19 (Actual); Study Completion 2015-08-19 (Actual)

PRIMARY OUTCOMES:
Safety of hESC derived RPE cells | 12 Months
  The transplantation of hESC-derived RPE cells MA09-hRPE will be considered safe and tolerated in the absence of:
  * Any grade 2 (NCI grading system) or greater adverse event related to the cell product
  * Any evidence that the cells are contaminated with an infectious agent
  * Any evidence that the cells show tumorigenic potential

SECONDARY OUTCOMES:
exploratory evaluations for potential efficacy endpoints. | 12 months
  Secondary endpoints will be evaluated as exploratory evaluations for potential efficacy endpoints.
  * Change in the mean of BCVA
  * Autofluorescence photography
  * Reading speed
  Evidence of successful engraftment will consist of:
  * Structural evidence (OCT imaging, fluorescein angiography, slit-lamp examination with fundus photography) that cells have been implanted in the correct location
  * Electroretinographic evidence (mfERG) showing enhanced activity in the implant location

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (4):
- United States (4):
  - Jules Stein Eye Institute, UCLA School of Medicine, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Mass Eye and Ear, Boston, Massachusetts
  - Wills Eye Institute-Mid Atlantic Retina, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Schwartz SD, Regillo CD, Lam BL, Eliott D, Rosenfeld PJ, Gregori NZ, Hubschman JP, Davis JL, Heilwell G, Spirn M, Maguire J, Gay R, Bateman J, Ostrick RM, Morris D, Vincent M, Anglade E, Del Priore LV, Lanza R. Human embryonic stem cell-derived retinal pigment epithelium in patients with age-related macular degeneration and Stargardt's macular dystrophy: follow-up of two open-label phase 1/2 studies. Lancet. 2015 Feb 7;385(9967):509-16. doi: 10.1016/S0140-6736(14)61376-3. Epub 2014 Oct 15. PMID 25458728
- [Derived] Schwartz SD, Hubschman JP, Heilwell G, Franco-Cardenas V, Pan CK, Ostrick RM, Mickunas E, Gay R, Klimanskaya I, Lanza R. Embryonic stem cell trials for macular degeneration: a preliminary report. Lancet. 2012 Feb 25;379(9817):713-20. doi: 10.1016/S0140-6736(12)60028-2. Epub 2012 Jan 24. PMID 22281388
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;7316-CL-0002
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217491&parentIdentifier=7316-CL-0002&attachmentIdentifier=969e8c99-a995-4b49-814d-8c62522cafbe&fileName=7316-CL-0002_0005_Plain_language_summary.pdf&versionIdentifier=